CLINICAL TRIAL: NCT00888446
Title: Phase II, Placebo-controlled, Double-blind, Dose-escalation/Dose-optimization Trial to Evaluate Safety and Immunogenicity of tgAAC09, an HIV Vaccine Containing Clade C Gag-PR-ΔRT DNA in an Adeno-associated Virus (AAV) Capsid
Brief Title: Safety and Immunogenicity Study of tgAAC09, an HIV Vaccine in an Adeno-associated Virus (AAV) Capsid
Acronym: TGC14F
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Targeted Genetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IAVI A002
Record Dates: First submitted 2009-04-23; First posted 2009-04-27 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Human Immunodeficiency Virus Infections; HIV Infections
Keywords: HIV; HIV seronegativity; preventative vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Group A (Experimental): Number of Vaccine Recipients: 10
  Dosage level 3 x 10^10 DRP
  Month 0 + 6
  Interventions: Biological: tgAAC09
- Group B (Experimental): Number of Vaccine Recipients: 10
  Dosage level 3 x 10^10 DRP
  Month 0+12
  Interventions: Biological: tgAAC09
- Group C (Experimental): Number of Vaccine Recipients: 10
  Dosage level 3 x 10^11 DRP
  Month 0+6
  Interventions: Biological: tgAAC09
- Group D (Experimental): Number of Vaccine Recipients: 10
  Dosage level 3 x 10^11 DRP
  Month 0+12
  Interventions: Biological: tgAAC09
- Group E (Experimental): Number of Vaccine Recipients: 10
  Dosage level 3 x 10^12 DRP
  Month 0+6
  Interventions: Biological: tgAAC09
- Group F (Experimental): Number of Vaccine Recipients: 10
  Dosage level 3 x 10^12 DRP
  Month 0+12
  Interventions: Biological: tgAAC09
- Group G (Experimental): Number of Vaccine Recipients: 10
  Preselected for baseline AAV neutralization titers of <1/8
  Dosage level 3 x 10^12 DRP
  Month 0+6
  Interventions: Biological: tgAAC09
- Placebo (Placebo Comparator): 3 volunteers will receive placebo matched to each experimental group.
  Interventions: Other: Formulation buffer

INTERVENTIONS:
Biological: tgAAC09
  Arms: Group A; Group B
Biological: tgAAC09
  Arms: Group C; Group D
Biological: tgAAC09
  Arms: Group E; Group F; Group G
Other: Formulation buffer — Sterile isotonic buffered salt solution
  Arms: Placebo

SUMMARY:
This phase 2 study will evaluate the safety, immunogenicity and optimal timing of two injections at three dose levels of the tgAAC09 vaccine in healthy volunteers. Study volunteers will receive two intramuscular injections of tgAAC09 or placebo at Months 0 and 6 (groups A, C, E and G) or at Months 0 and 12 (groups B, D and F) and be followed for a total of 18 months following the first injection with the exception of group G in which volunteers will be followed for 12 months after the first injection (6 months after the second injection). This study will explore whether boosting is possible, and compare a shorter and more practical six-month time interval with a twelve-month time interval.

DETAILED DESCRIPTION:
The study design will also assess the effect of the presence of anti-AAV2 capsid neutralizing antibodies at the time of vaccination on the safety and immunogenicity of tgAAC09. Since the prevalence of pre-existing neutralizing antibodies to AAV2 capsid is high (IAVI and Targeted Genetics, data on file), this protocol amendment adds Group G which is composed of volunteers who have documented pre-existing anti-AAV2 capsid neutralizing antibodies titers ≤ 1/8. This will assure that there are sufficient numbers of volunteers with and without antibodies for a useful comparison.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Age at least 18 years on the day of screening and no greater than 50 years on the day of the first study injection
* Willing to comply with the requirements of the protocol and available for follow up for the planned duration of the study
* Able and willing to give informed consent.
* Willing to undergo HIV testing, counseling and receive results
* If sexually active female of child-bearing potential (not menopausal or anatomically sterile), willing to use an effective method of contraception (hormonal contraceptives; intrauterine contraceptive device (IUCD); condoms; anatomical sterility in self or partner) from screening until at least four months after last study injection and willing to undergo urine pregnancy tests at screening, prior to each injection and four months after the last injection
* If sexually active male, willing to use a method of contraception (such as condoms) from screening until four months after the last study injection

Exclusion Criteria:

* HIV-1 or HIV-2 infection
* Active tuberculosis
* Clinically relevant abnormality on history or examination including history of immunodeficiency, or cancer, or autoimmune disorder
* Use of systemic corticosteroids, immunosuppressive or anticancer medications in the last six months
* Chronic condition that, in the opinion of the investigator or the designated trial physician, would make the volunteer unsuitable for the study
* Any of the following abnormal laboratory parameters:

  * Hemoglobin <9.0 g/dL (females), <12.0 g/dL (males)
  * Absolute Neutrophil Count (ANC): ≤ 999/mm3
  * Absolute Lymphocyte Count (ALC): ≤ 500/mm3
  * Platelets: decreased ≤ 90,000 or increased ≥ 550,000/mm3
  * Creatinine: > 1.4 x ULN
  * AST: >3.0 x ULN
  * ALT: >3.0 x ULN
  * Urine dipstick: blood = 2+ or more (except in menstruating females); protein = 2+ or more
* Any of the following high-risk behaviors:

  * Had unprotected vaginal or anal sex with a known HIV positive person in the past six months
  * Had unprotected vaginal or anal sex with a casual partner (i.e. no continuing established relationship) in the past six months
  * Engaged in sex work for money or drugs in the past six months
  * Used injection drugs illegally in the past six months
  * Acquired a sexually transmitted infection (STI) in the past six months
* If female, pregnant, lactating or planning a pregnancy within four months after last study injection
* Receipt of live attenuated vaccine within 30 days or other vaccine within 14 days of the first study injection
* Receipt of blood transfusion or blood products six months prior to the first study injection
* Participation in another clinical trial of an investigational product currently or within last 12 weeks of first study injection or expected participation during this study
* Prior receipt of an investigational HIV vaccine
* History of severe local or systemic reaction to vaccination(s) or history of severe allergic reactions
* History of major neurological or psychiatric disorders
* Positive for hepatitis B surface antigen, active untreated syphilis (confirmed by treponemal test such as TPHA in addition to nontreponemal test such as RPR) or other active sexually transmitted diseases

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Safety: proportion of volunteers with severe local and systemic reactions, proportion of volunteers with other SAEs (including laboratory abnormalities) related to study vaccine, number of volunteers with SAEs related to study vaccine | 18 months
Proportion of volunteers with HIV-1 specific T- cell responses quantified by γ-IFN ELISPOT and magnitude of the response, and proportion of volunteers with HIV-1 specific binding antibodies and magnitude of the response | 18 months

SECONDARY OUTCOMES:
Safety: high versus low or negative titres of neutralizing antibodies to AAV2 at the time of each vaccination | 18 months
Immunogenicity: proportion of volunteers with HIV-1 specific T- cell responses by γ-IFN CFC or other T-cell assays | 18 months
Immunogenicity endpoints in volunteers with high versus low or negative titres of neutralizing antibodies to AAV2 at the time of each vaccination | 18 months
Immunogenicity endpoints in volunteers with versus without four-fold or greater increase in titres of neutralizing antibodies to AAV2 after vaccination | 18 months
Immunogenicity endpoints after the second study injection, compared with the first study injection | 18 months
Immunogenicity endpoints after the second study injection following a twelve-month interval compared to a six-month interval | 18 months
Vaccine biodistribution: presence and persistence of vaccine in peripheral blood mononuclear cells (PBMC), saliva, nasal swabs, urine and semen or cervical/vaginal secretions | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Eftyhia Vardas, MD, Study Chair — Perinatal HIV Research Unit (PHRU), Baragwanath; Linda-Gail Bekker, MD, Principal Investigator — Desmond Tutu HIV Centre Cape Town; Anwar Hoosen, Principal Investigator — Medical University of Southern Africa (Medunsa); Elwyn Chomba, MD, Principal Investigator — Zambia-Emory HIV Research Project (ZEHRP), Lusaka; Pontiano Kaleebu, MD, PhD, Principal Investigator — MRC/UVRI and LSHTM Uganda Research Unit
Locations (5):
- South Africa (3):
  - Desmond Tutu HIV Centre Cape Town, Cape Town, South Africa
  - Medunsa, South Africa, South Africa
  - Perinatal HIV Research Unit, Baragwanath Hospital, Soweto, South Africa
- Uganda Virus Research Institute, Entebbe, Entebbe, Uganda
- Zambia-Emory HIV Research Project (ZEHRP), Lusaka, Lusaka Province, Zambia

REFERENCES:
- [Result] Vardas E, Kaleebu P, Bekker LG, Hoosen A, Chomba E, Johnson PR, Anklesaria P, Birungi J, Barin B, Boaz M, Cox J, Lehrman J, Stevens G, Gilmour J, Tarragona T, Hayes P, Lowenbein S, Kizito E, Fast P, Heald AE, Schmidt C. A phase 2 study to evaluate the safety and immunogenicity of a recombinant HIV type 1 vaccine based on adeno-associated virus. AIDS Res Hum Retroviruses. 2010 Aug;26(8):933-42. doi: 10.1089/aid.2009.0242. PMID 20666584
- See also: Related Info — http://www.iavi.org